CLINICAL TRIAL: NCT06429267
Title: Comprehensive Investigation of Bioabsorbable Screws in Pediatric Orthopedic Surgery: Mechanical Properties, Long-term Performance, and Practical Applications
Brief Title: Investigation Of Bioabsorbable Screws In Pediatric Orthopedic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6360
Record Dates: First submitted 2024-05-01; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Pediatric; Fracture; Orthopedic Devices Associated With Misadventures, Surgical Instruments, Materials and Devices (Including Sutures); Patient Satisfaction
MeSH Terms: conditions — Fractures, Bone; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two groups which will determine the type of screw (stainless steel or bioabsorbable) in their surgery.
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control Group (Receiving Metal Screws) (Active Comparator): Patients that are randomly assigned to receive traditional, metal screws
  Interventions: Device: Metal/Titanium Screw
- Experimental Group (Receiving Bioabsorbable Screws) (Experimental): Patients that are randomly assigned to receive Bioabsorbable screws
  Interventions: Device: Bioabsorbable Screw

INTERVENTIONS:
Device: Bioabsorbable Screw — Bioabsorbable screw that redissolves into the bone. Mineral fibers are composed of Silicon Dioxide (SiO2), Sodium Oxide, Calcium Oxide, Magnesium Oxide, Boron Trioxide, and Phosphorous Pentoxide
  Other Names: Ossiofiber
  Arms: Experimental Group (Receiving Bioabsorbable Screws)
Device: Metal/Titanium Screw — Traditional metal screw used in fracture fixation that requires hardware removal
  Other Names: OrthoPediatrics
  Arms: Control Group (Receiving Metal Screws)

SUMMARY:
This study is a prospective randomized controlled trial comparing the clinical outcomes of bioabsorbable screws to conventional metal screws in pediatric patients (aged 0 to 18) undergoing surgical fixation for trauma or elective procedures. Conducted by the pediatric orthopedic department at Children's Hospital New Orleans, the study aims to evaluate the effectiveness of these screws in bone healing over key post-operative intervals (6 weeks, 6 months, and 1 year). It seeks to determine if bioabsorbable screws offer significant advantages over metal screws in terms of reducing the need for secondary surgeries, based on their hypothesized noninferiority in complication rates. Participants will be randomly assigned to receive either bioabsorbable or metal (titanium or stainless steel) screws after obtaining informed consent from a parent or guardian.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled trial to evaluate clinical outcomes associated with the use of bioabsorbable screws compared to conventional metal screws in children aged 0 to 18 who are undergoing surgical fixation in the setting of trauma such as medial epicondyle fractures of the elbow or elective procedures. The research will be conducted within the pediatric orthopedic department at CHNOLA, and participants will be assessed at key intervals, including 6 weeks, 6 months, and 1 year post-operation post-operation. The primary objective of this study is to assess and compare the effectiveness of conventional metal screws and bioabsorbable screws in bone healing. This study aims to determine whether bioabsorbable screws are significantly superior to conventional titanium screws. The investigators hypothesize bioabsorbable screws are significantly noninferior to conventional metal screws in terms of complications based on prior surgical constructs that demonstrate bioabsorbable screws eliminate the need for a second surgery After informed consent has been obtained from the parents of patients, eligible patients undergoing cannulated screw fixation will be randomized into two groups: one group who will receive bioabsorbable screws and the other group who will receive metal screws (titanium or stainless steel).

ELIGIBILITY:
Inclusion Criteria:

* Primary fractures requiring fixation with cannulated screws

Exclusion Criteria:

* Children ten years old or under with a fracture requiring screws to be fixed across the growth plate (physis)
* Secondary fractures
* Non-union fractures
* Tibial tubercle osteotomies (TTOs)
* Slipped capital femoral epiphysis (SCFEs)
* Unable or unwilling to provide informed consent or parental/guardian consent for participants under 18 years of age
* Allergies or contraindications to screw materials

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Computer Adaptive PROMIS (Patient-Reported Outcomes Measurement Information System) Surveys | 6 weeks, 6 months, 1 year
  Pain, Upper Extremity and Mobility. These questionnaires are scored using T scores. For pain, a higher score is a worse outcome. For mobility and upper extremity, a lower score is a worse outcome. Min value is 0 and max is 100 for all.

SECONDARY OUTCOMES:
Complications | 1 year
  Any complications of surgery (infection etc)

CONTACTS AND LOCATIONS:
Overall Officials: Carter Clement, MD, MBA, Principal Investigator — LSUHSC
Locations (1):
- Children's Hospital New Orleans, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication